CLINICAL TRIAL: NCT04343170
Title: Effect of Ultra-short-term Treatment of Patients With Iron Deficiency or Anemia Undergoing Adolescent Scoliosis Correction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amany Faheem, Principal Investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ultrashort treatment of anemia
Record Dates: First submitted 2020-04-03; First posted 2020-04-13 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Ultra-short-term; Iron Deficiency Anemia; Scoliosis Idiopathic
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferric carboxymaltose; Vitamin B 12; Folic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Placebo Comparator): Patients of this group received placebo treatment consisted of two subcutaneous injections of 1 mL saline and an oral placebo.
  Interventions: Drug: Placebo
- ultra-short-term treatment (Experimental): Patients of this group received Combination treatment consisted of a slow (30 min) intravenous infusion of 20 mg/kg ferric carboxymaltose (maximum of 1000 mg), 40 000 U subcutaneous α erythropoietin,1 mg subcutaneous vitamin B12(, and 5 mg oral folic acid (acidum folicum)
  Interventions: Drug: ferric carboxymaltose , α erythropoietin, vitamin B12, oral folic acid

INTERVENTIONS:
Drug: Placebo — Patients of this group received placebo treatment consisted of two subcutaneous injections of 1 mL saline and an oral placebo
  Arms: control group
Drug: ferric carboxymaltose , α erythropoietin, vitamin B12, oral folic acid — Patients of this group received Combination treatment consisted of a slow (30 min) intravenous infusion of 20 mg/kg ferric carboxymaltose (maximum of 1000 mg), 40 000 U subcutaneous α erythropoietin,1 mg subcutaneous vitamin B12(, and 5 mg oral folic acid (acidum folicum)
  Arms: ultra-short-term treatment

SUMMARY:
Scoliosis is a condition in which there is curvature of the spine occurring in the lateral plane. It occurs in structural forms, characterized by a fixed curve, and "functional" forms, characterized by a flexible or correctable curve. By anatomic necessity, this lateral deviation is associated with vertebral rotation, such that when this deformity occurs in the thoracic spine, a chest wall deformity, or "rib hump," develops.

Often there is a primary structural curve with an adjacent secondary compensatory curve. Most cases of structural scoliosis are idiopathic and have their onset in early adolescence. Females are affected more often than males, and their curvature is more likely to worsen.

Lumbar fusion surgery is usually associated with massive blood loss. In clinical practice the surgeon might measure the visible peri-operative bleeding including intra- and post-operative drainage, but ignore blood component penetration into the tissues, residual blood in vertebral canal and loss due to haemolysis, which are also known as hidden blood loss.

In patients with adolescent idiopathic scoliosis (AIS), surgical treatment involves a posterior approach with multi-segmental pedicle screw fixation. Although this procedure is generally considered safe with few surgical complications, there are considerable variations in fusion length, surgical time, and the extent of soft-tissue exposure. Consequently, perioperative blood loss can be substantial, and the use of intraoperative and postoperative RBC transfusions are frequently required.

Patient blood management (PBM) is an evidence-based, multidisciplinary approach developed over the last 10 years focusing on improving patient outcomes as well as reducing the use of RBC transfusions. PBM includes several preventive measures to manage bleeding risks, reduce iatrogenic blood loss, and modify decision thresholds for the appropriate administration of blood therapy.

All patients for elective surgery in whom blood loss is expected to be > 500 ml should have their hemoglobin checked pre-operatively and be investigated if they are found to be anemic. In the general population, anemia is defined as a hemoglobin less than 130 g. in men and less than 120g. in women by the WHO. It was proposed that the cut-off value/trigger be changed to hemoglobin more than 130 g for both men and women. Women with hemoglobin levels between 120 and 129 g. are not considered to be anemic according to the WHO definition, leaving them at a potential disadvantage when undergoing major surgery

DETAILED DESCRIPTION:
44 Patients will be randomly classified into two equal groups each of 22 patients Group I: Patients of this group received Combination treatment consisted of a slow (30 min) intravenous infusion of 20 mg/kg ferric carboxymaltose (maximum of 1000 mg), 40 000 U subcutaneous α erythropoietin,1 mg subcutaneous vitamin B12(, and 5 mg oral folic acid (acidum folicum) Group II: Patients of this group received placebo treatment consisted of two subcutaneous injections of 1 mL saline and an oral placebo. Either iron or placebo (0•9% saline) were given intravenously via a black infusion set from behind a screen to assure blinding of the patient by a person not involved in data capturing or data entering.

Patient's vital signs will be monitored during and at least 15 min after drug application. Treatment will be given one day before the operation

Measurements:

1. Demographic data
2. The number of RBC transfusions during the first 7 days.
3. Perioperative course of Hb, (reticulocyte count, reticulocyte Hb content).
4. The need of fresh frozen plasma units transfused in first 7 days
5. The need of platelets units transfused in first 7 days
6. Platelet count.
7. Total leucocyte counts.
8. International normalized ratio.
9. Serum creatinine.
10. C-reactive protein,
11. Calculated RBC loss (preoperative RBC mass minus RBC mass at postoperative fifth day plus transfused RBC mass)
12. Length of ICU stay.
13. Incidence of acute kidney injury
14. Infections requiring antibiotics

ELIGIBILITY:
Inclusion Criteria:

* patients with idiopathic adolescent scoliosis
* patients with anemia (haemoglobin concentration (Hb) <12g/dL in women and Hb <13 g/dL in men)
* patients with isolated iron deficiency (ferritin <100 mcg/L, no anemia)

Exclusion Criteria:

1. Impairments, diseases (renal &/ hepatic) or language problems which do not allow the patient to fully understand the consequences of study participation
2. Known allergy against iron - carboxymaltose
3. Hemoglobin concentration (Hb) <90 g/L in both male and female)

Ages: 13 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
percentage of patients not required blood transfusion | up to 7 days postoperative
  percentage of patients not required blood transfusion

SECONDARY OUTCOMES:
the length in I.C.U | during ICU stay period up to 7 days postoperative
  the length in I.C.U by days
the incidence of acute kidney injury | up to 7 days postoperative
  number of patients developed acute kidney injury
incidence of infections requiring antibiotic treatment | up to 7 days postoperative
  number of patients developed infections requiring antibiotic treatment
perioperative hemoglobin | up to 7 days postoperative
  perioperative hemoglobin by gm
perioperative platelet | up to 7 days postoperative
  perioperative platelet presented as platelet count per microliter of blood
perioperative leucocyte counts | up to 7 days postoperative
  perioperative leucocyte counts presented as white blood cells per microliter
calculated Red blood cells loss | up to 7 days postoperative
  calculated Red blood cells loss by ml

CONTACTS AND LOCATIONS:
Locations (1):
- tarek Abdel Lattif, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No